CLINICAL TRIAL: NCT01430286
Title: Evaluation of a Web-based Psycho-Educational Program for Informal Caregivers of Patients With Alzheimer's Disease (AD).
Brief Title: Web-based Psycho-Educational Program to Support Carers of Alzheimer's Patients
Acronym: DIAPASON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Direction de l'Hospitalisation et de l'Organisation des Soins (PREQHOS) (Unknown); Fondation Mederic Alzheimer (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P081002
Record Dates: First submitted 2011-08-22; First posted 2011-09-08 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
Keywords: Caregivers; Alzheimer Disease; Psychological stress; Psychological adaptation; Self-efficacy; Randomized controlled trial
MeSH Terms: conditions — Alzheimer Disease; Stress, Psychological | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psycho-educational program (Experimental): This group is trained for a 3 month period by a web-based psycho-educational program, Lifestyle Counseling, etc.
  Interventions: Behavioral: psycho-social intervention based on a web-based psycho-educational program, called Diapason.
- Standard treatment (Active Comparator): This group will receive treatment as usual : consultation in memory clinic every 6 months during the AD patient's consultation.
  Interventions: Behavioral: Consultation in memory clinic

INTERVENTIONS:
Behavioral: psycho-social intervention based on a web-based psycho-educational program, called Diapason. — This group will be trained for a 3 month period by a web-based psycho-educational program, Lifestyle Counseling, etc.
  Other Names: Web-based psycho-educational program
  Arms: Psycho-educational program
Behavioral: Consultation in memory clinic — This group will receive treatment as usual (consultation in memory clinic every 6 months)
  Arms: Standard treatment

SUMMARY:
The aim of the project is to evaluate the efficacy of a web-based psycho-educational programme designed to support informal caregivers of patients with Alzheimer's disease (AD).This program focuses on information about the illness, her progression, how to prevent psychological strain using anticipation and relaxation techniques and providing a virtual space (forum) to discuss with other caregivers.

DETAILED DESCRIPTION:
Context: Since some of the ICs do not have the possibility to participate in face-to-face interventions, information and communication technologies are being increasingly used for a distance intervention. Research showing the benefit of a combined approach including psycho-social interventions for caregivers and Information and Communication Technologies (ICT) in the caring of Alzheimer's disease patients is actually growing. Main objective: To evaluate the efficacy of a a web-based psycho-educational program designed to support carers of AD patientsMethodology: This is a randomized clinical trial . 80 participants will be randomized in 2 parallel groups: The volunteers in the experimental condition (EC) should visit at least one time per week the website of program, during 12 weeks. Each week a new thematic is added to the website. b) The participants in the control group (CG) will receive a minimal intervention, and will have access to the Diapason program after their participation (six months). Caregivers are recruited (according to exclusion and inclusion criteria) and followed up in memory center participating in the trial.

Evaluation criteria:

Primary criteria:

- Perceived Stress Scale (PSS-14).

Secondary evaluation criteria:

* Nottingham Health Profile (NPH),
* Zarit Burden Interview (BI),
* Revised Memory and Behavior Problems Checklist (RMBPC),
* Beck Depression Inventory (BDI-2) Mediator variables
* Revised Scale for Caregiving Self-Efficacy (RCSE).
* Statistics of website utilization Controlled variables
* Sociodemographic variables (Self report)
* Knowledge about illness (Visual analogical scale - VAS)
* The quality of the relationship with the patient (VAS)
* Time spent on caregiving
* Other sources of stress (i.e. work, health status, financial status)
* Respite or social help (i.e. psychotherapy, associations, technical help, etc)
* Cognitive and autonomy status of patient (MMSE and IADL)

Statistical analysis by the department of biostatistics and medical computing of the Hospital Cochin will be performed.

ELIGIBILITY:
Inclusion criteria :

* Family caregivers of AD patients DSM IV-TR (American Psychiatric Association 2004) or NINCDS/ADRDA (McKhann et al. 1984).
* Age: over 18 years old
* score 12 or over on the Perceived Stress Scale 14 items (PSS-14, Cohen) Need for information or help
* Sign informed consent

Exclusion criteria :

* Professional or paid caregiver
* Physical or mental disease incompatible with patient's management
* Impossibility to participate in the educational program
* Absence of perceived stress
* Ongoing psychotherapy or a similar program in parallel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Perceived stress | every 3 months (between 0 and 6 months)
  Stress perceived by the caregiver is measured by the French version of the Perceived Stress Scale, the version of 14 items from Cohen and colleagues (1983), traduced to by Bruchon-Schweitzer in 2002. The PSS-14 is a widely used self-reported scale, evaluating the general appraisal of stress in the last month. It consists in 14 items, which scores range from 0 (never) to 4 (very often). This scale has demonstrated a high reliability and validity in several studies. The total score range is 0-56. In this study CG and EC will perform the scale at baseline (month 0), at the end of intervention for EC (month 3) and follow-up (month 6). Participants from control group will receive an acces to the program at the end of the last visit (M6).

SECONDARY OUTCOMES:
Nottingham Health Profile (NPH) | every 3 months (between 0 and 6 months)
ZARIT Burden Interview (BI) | every 3 months (between 0 and 6 months)
Revised Memory and Behavior Problems Checklist (RMBPC) | every 3 months (between 0 and 6 months)
Beck Depression Inventory (BDI-2) | every 3 months (between 0 and 6 months)
Revised Scale for Caregiving Self-Efficacy (RCSE) | every 3 months (between 0 and 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Rigaud, MD, PhD, Principal Investigator — Hôpital Broca - la Collégiale, Memory Clinic
Locations (1):
- Hôpital Broca - la Collégiale, Geriatric Unit, Memory Clinic, Paris, France

REFERENCES:
- [Background] Ankri J, Andrieu S, Beaufils B, Grand A, Henrard JC. Beyond the global score of the Zarit Burden Interview: useful dimensions for clinicians. Int J Geriatr Psychiatry. 2005 Mar;20(3):254-60. doi: 10.1002/gps.1275. PMID 15717336
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Bourgeois MS, Schulz R, Burgio L. Interventions for caregivers of patients with Alzheimer's disease: a review and analysis of content, process, and outcomes. Int J Aging Hum Dev. 1996;43(1):35-92. doi: 10.2190/AN6L-6QBQ-76G0-0N9A. PMID 8886875
- [Background] Brodaty H, Green A, Koschera A. Meta-analysis of psychosocial interventions for caregivers of people with dementia. J Am Geriatr Soc. 2003 May;51(5):657-64. doi: 10.1034/j.1600-0579.2003.00210.x. PMID 12752841
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] Eisdorfer C, Czaja SJ, Loewenstein DA, Rubert MP, Arguelles S, Mitrani VB, Szapocznik J. The effect of a family therapy and technology-based intervention on caregiver depression. Gerontologist. 2003 Aug;43(4):521-31. doi: 10.1093/geront/43.4.521. PMID 12937331
- [Background] Gallagher-Thompson D, Coon DW. Evidence-based psychological treatments for distress in family caregivers of older adults. Psychol Aging. 2007 Mar;22(1):37-51. doi: 10.1037/0882-7974.22.1.37. PMID 17385981
- [Background] Gottlieb BH, Wolfe J. Coping with family caregiving to persons with dementia: a critical review. Aging Ment Health. 2002 Nov;6(4):325-42. doi: 10.1080/1360786021000006947. PMID 12425767
- [Background] Livingston G, Manela M, Katona C. Depression and other psychiatric morbidity in carers of elderly people living at home. BMJ. 1996 Jan 20;312(7024):153-6. doi: 10.1136/bmj.312.7024.153. PMID 8563534
- [Background] Lyketsos CG, Steinberg M, Tschanz JT, Norton MC, Steffens DC, Breitner JC. Mental and behavioral disturbances in dementia: findings from the Cache County Study on Memory in Aging. Am J Psychiatry. 2000 May;157(5):708-14. doi: 10.1176/appi.ajp.157.5.708. PMID 10784462
- [Background] McKhann G, Drachman D, Folstein M, Katzman R, Price D, Stadlan EM. Clinical diagnosis of Alzheimer's disease: report of the NINCDS-ADRDA Work Group under the auspices of Department of Health and Human Services Task Force on Alzheimer's Disease. Neurology. 1984 Jul;34(7):939-44. doi: 10.1212/wnl.34.7.939. PMID 6610841
- [Background] Mahoney DF, Tarlow BJ, Jones RN. Effects of an automated telephone support system on caregiver burden and anxiety: findings from the REACH for TLC intervention study. Gerontologist. 2003 Aug;43(4):556-67. doi: 10.1093/geront/43.4.556. PMID 12937334
- [Background] Magnusson L, Hanson E, Brito L, Berthold H, Chambers M, Daly T. Supporting family carers through the use of information and communication technology--the EU project ACTION. Int J Nurs Stud. 2002 May;39(4):369-81. doi: 10.1016/s0020-7489(01)00034-7. PMID 11909614
- [Background] Mittelman MS, Roth DL, Haley WE, Zarit SH. Effects of a caregiver intervention on negative caregiver appraisals of behavior problems in patients with Alzheimer's disease: results of a randomized trial. J Gerontol B Psychol Sci Soc Sci. 2004 Jan;59(1):P27-34. doi: 10.1093/geronb/59.1.p27. PMID 14722336
- [Background] Moniz-Cook E, Vernooij-Dassen M, Woods R, Verhey F, Chattat R, De Vugt M, Mountain G, O'Connell M, Harrison J, Vasse E, Droes RM, Orrell M; INTERDEM group. A European consensus on outcome measures for psychosocial intervention research in dementia care. Aging Ment Health. 2008 Jan;12(1):14-29. doi: 10.1080/13607860801919850. PMID 18297476
- [Background] Ramaroson H, Helmer C, Barberger-Gateau P, Letenneur L, Dartigues JF; PAQUID. [Prevalence of dementia and Alzheimer's disease among subjects aged 75 years or over: updated results of the PAQUID cohort]. Rev Neurol (Paris). 2003 Apr;159(4):405-11. French. PMID 12773869
- [Background] Schulz R, O'Brien AT, Bookwala J, Fleissner K. Psychiatric and physical morbidity effects of dementia caregiving: prevalence, correlates, and causes. Gerontologist. 1995 Dec;35(6):771-91. doi: 10.1093/geront/35.6.771. PMID 8557205
- [Background] Schulz R, Beach SR. Caregiving as a risk factor for mortality: the Caregiver Health Effects Study. JAMA. 1999 Dec 15;282(23):2215-9. doi: 10.1001/jama.282.23.2215. PMID 10605972
- [Background] Schulz R, Martire LM, Klinger JN. Evidence-based caregiver interventions in geriatric psychiatry. Psychiatr Clin North Am. 2005 Dec;28(4):1007-38, x. doi: 10.1016/j.psc.2005.09.003. No abstract available. PMID 16325738
- [Background] Sorensen S, Pinquart M, Duberstein P. How effective are interventions with caregivers? An updated meta-analysis. Gerontologist. 2002 Jun;42(3):356-72. doi: 10.1093/geront/42.3.356. PMID 12040138
- [Background] Teri L. Behavior and caregiver burden: behavioral problems in patients with Alzheimer disease and its association with caregiver distress. Alzheimer Dis Assoc Disord. 1997;11 Suppl 4:S35-8. PMID 9339271
- [Background] Teri L, Logsdon RG, McCurry SM. Nonpharmacologic treatment of behavioral disturbance in dementia. Med Clin North Am. 2002 May;86(3):641-56, viii. doi: 10.1016/s0025-7125(02)00006-8. PMID 12168563
- [Background] Yesavage JA. Geriatric depression scale: consistency of depressive symptoms over time. Percept Mot Skills. 1991 Dec;73(3 Pt 1):1032. doi: 10.2466/pms.1991.73.3.1032. No abstract available. PMID 1792116
- [Background] Zarit SH, Todd PA, Zarit JM. Subjective burden of husbands and wives as caregivers: a longitudinal study. Gerontologist. 1986 Jun;26(3):260-6. doi: 10.1093/geront/26.3.260. No abstract available. PMID 3721233
- [Background] Cristancho-Lacroix V, Moulin F, Wrobel J, Batrancourt B, Plichart M, De Rotrou J, Cantegreil-Kallen I, Rigaud AS. A web-based program for informal caregivers of persons with Alzheimer's disease: an iterative user-centered design. JMIR Res Protoc. 2014 Sep 15;3(3):e46. doi: 10.2196/resprot.3607. PMID 25263541
- [Background] Cristancho-Lacroix V, Wrobel J, Cantegreil-Kallen I, Dub T, Rouquette A, Rigaud AS. A web-based psychoeducational program for informal caregivers of patients with Alzheimer's disease: a pilot randomized controlled trial. J Med Internet Res. 2015 May 12;17(5):e117. doi: 10.2196/jmir.3717. PMID 25967983
- [Background] Cristancho-Lacroix V, Kerherve H, de Rotrou J, Rouquette A, Legouverneur G, Rigaud AS. Evaluating the efficacy of a web-based program (diapason) for informal caregivers of patients with Alzheimer's disease: protocol for a randomized clinical trial. JMIR Res Protoc. 2013 Dec 6;2(2):e55. doi: 10.2196/resprot.2978. PMID 24317497
- [Derived] Gonzalez-Fraile E, Ballesteros J, Rueda JR, Santos-Zorrozua B, Sola I, McCleery J. Remotely delivered information, training and support for informal caregivers of people with dementia. Cochrane Database Syst Rev. 2021 Jan 4;1(1):CD006440. doi: 10.1002/14651858.CD006440.pub3. PMID 33417236